CLINICAL TRIAL: NCT02607241
Title: Comparison of a Paclitaxel-Coated Balloon Without Stent Implantation Against a Drug-Eluting Bioresorbable Scaffold for Treatment of Stable Coronary Artery Disease: A Prospective Randomized Study Using Optical Coherence Tomography
Brief Title: Comparison of Paclitaxel-Coated Balloons Against Drug-Eluting Bioresorbable Scaffolds for Elective PCI Using OCT
Acronym: OCTOPUS-3
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The product used in the comparator arm (BRS) has become unavailable in April 2017. The recruitment has been stopped.
Sponsor: University of Jena (Other)
Collaborators: KKS Netzwerk (Network)
Responsible Party: Principal Investigator, Tudor C. Poerner, MD, PD Dr. med. Tudor C. Poerner, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKJ-TCP-3
Record Dates: First submitted 2015-11-15; First posted 2015-11-18 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Coronary Artery Disease
Keywords: drug-coated balloon; bioresorbable scaffold; fractional flow reserve; optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BRS (Active Comparator): OCT-guided BRS implantation: implantation of a bioresorbable scaffold (BRS) under OCT guidance.
  Note: Absorb™ from Abbott Vascular has been used as BRS until this product became unavailable in April 2017. Currently the recruitment is stopped due to this issue, until the use of another BRS gets final approval.
  Interventions: Device: OCT-guided BRS implantation
- DCB-only (Experimental): FFR-guided DCB-only PCI: PCI using DCB (SeQuent Please™, B Braun Melsungen GmBH) without stent implantation und FFR guidance
  Interventions: Device: FFR-guided DCB-only PCI

INTERVENTIONS:
Device: OCT-guided BRS implantation — Implantation of a BRS using OCT to measure vessel size, choose BRS size and length and assess implantation results and the need of further postdilations
  Arms: BRS
Device: FFR-guided DCB-only PCI — PCI performed under FFR guidance using following algorithm: (1) predilation followed by angiographic assessment of residual stenosis and dissections; (2) evaluate suitability for DCB-only, which is deemed feasible if the FFR > 0.8, residual diameter stenosis < 40% and no flow-limiting dissections are observed; (3) DCB dilation and (4) assessment of final results using FFR and QCA measurements. Provisional stenting is allowed only if the final PCI results are not acceptable (flow-limiting dissection, residual stenosis > 40% or FFR < 0.8).
  Arms: DCB-only

SUMMARY:
This prospective randomized clinical trial aims to compare two different "metal-free" strategies for elective percutaneous coronary revascularization: the FFR-guided DCB-only PCI (drug-coated balloon: SeQuent Please™, B Braun Melsungen GmBH) vs. OCT-guided BRS implantation (bioresorbable scaffold: Absorb™, Abbott Vascular).

DETAILED DESCRIPTION:
Background:

Coronary artery disease (CAD) accounts for most deaths in the industrialized countries due to its high prevalence of 6-8%. CAD is mainly treated by percutaneous coronary interventions (PCI), which currently involve in over 90% of cases the implantation of metallic stents, mostly as drug-eluting devices(DES). Despite continuous technological advancement over the last decade, DES are still limited at long-term follow-up by restenosis and also by the risk of thrombosis, occurring in 5-20% and respectively 0.5-1.7% of cases. Therefore, two metal-free strategies are evaluated in order to overcome these intrinsic limitations of DES:

1. Bioresorbable scaffolds (BRS) proved comparable safety and efficacy at 1 year compared to best-in-class DES comparators and also showed in small substudies very promising 5-year results with restoration of vasomotricity and positive vessel remodeling. Optical coherence tomography (OCT) is the new gold standard for endovascular imaging of stents, atherosclerosis progression, vulnerable plaque and neointimal proliferation. OCT is currently recommended for both guidance of implantation and for assessment of long-term results of BRS.
2. Drug-coated balloons (DCB) were mainly employed to treat restenosis in metallic stents, but newer reports advocate their potential to be used as stand-alone treatment of de-novo stenoses without stenting, especially when fractional flow reserve (FFR) measurements are additionally used to assess PCI results.

This clinical trial evaluates the FFR-guided DCB-only (experimental arm: SeQuent Please™, B Braun Melsungen GmBH) PCI against the OCT-guided BRS implantation (comparator arm: Absorb™, Abbott Vascular) for treatment of stable CAD. The trial is designed as a non-inferiority, nationally conducted, multicenter, open-labeled, controlled study using a 1:1 block randomization and am invasive 6-9 month follow-up (f/u) by quantitative coronary angiography (QCA) and OCT.

Beyond the pre-specified endpoints the study mainly looking at suppression of neointimal proliferation, we will also investigate the patterns of healing and neointimal proliferation, the plaque morphology and neoatherosclerosis f/u using OCT at 6-9 months. Clinically, we attempt to record the major adverse cardiovascular events (MACE: acute myocardial infarction, cardiac death, TLR) up to 5 years after the index procedure.

A number of 196 patients scheduled for PCI with a native coronary stenosis suitable for BRS implantation and OCT imaging will be openly 1:1 randomized. This number of patients is considered to be sufficient to prove non-inferiority of DCB-only vs. BRS, using a margin of 0.2 mm with a confidence interval of 0.5 mm for the primary endpoint (diameter NLG).

ELIGIBILITY:
Inclusion Criteria:

* written consent
* indication for elective PCI of a de novo coronary stenosis in a native vessel
* coronary multivessel disease with clinically proven indication for repeating coronary angiography at 6-9 months (staged PCI strategy)

Exclusion Criteria:

* pregnancy, lactation, women of childbearing age w/o reliable contraception
* life expectance < 50 % at 1 year
* major surgery planned within 6 months
* participation in other clinical trials or impossibility to give written consent
* acute coronary syndrome or cardiogenic shock within the last 4 weeks
* stent thrombosis, defined as "probable" or "definite" by ARC
* contraindication against dual antiplatelet therapy
* allergy against mTOR-inhibitors or taxol derivates
* target lesion situated in the left main coronary artery, in a bypass graft or a grafted vessel
* reference luminal diameter of the target lesion > 3.75 mm or < 2.0 mm
* lesion length > 30 mm, bifurcation lesion requiring intervention on a major side branch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11; Primary Completion 2018-02 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Angiographic NLG | 6-9 months
  Absolute net luminal diameter gain measured by QCA as minimal luminal diameter at f/u - minimal luminal diameter at baseline within the region of interest

SECONDARY OUTCOMES:
Volumetric NLG | 6-9 months
  Absolute net luminal volumetric gain using three-dimensional OCT-based vessel segment reconstruction at f/u
Angiographic and volumetric LLL | 6-9 months
  Absolute late luminal diameter loss (LLL) using QCA and late luminal volumetric loss by OCT at f/u
TLR | 0-9 months
  % clinically driven target lesion revascularization (TLR) during f/u

OTHER OUTCOMES:
Acute TVF | 0-9 months
  Target vessel failure requiring emergent revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Tudor C Poerner, MD, Principal Investigator — Jena University Hospital
Locations (1):
- University Hospital of Jena, Heart Center, Division of Cardiology, Jena, Germany